CLINICAL TRIAL: NCT00793325
Title: Special Investigation Of Long Term Use Of Genotropin For SGA (Regulatory Post Marketing Commitment Plan)
Brief Title: Long Term Use of Somatropin in Patients Small for Gestational Age
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6281292
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-12

CONDITIONS: Small for Gestational Age
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Somatropin: Patients administered Somatropin.
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Genotropin® 5.3mg, Genotropin®inj.12mg, Genotropin®MiniQuick s.c. inj.0.6mg・1.0mg・1.4mg, depending on the Investigator prescription.
  Frequency and duration are according to Package Insert as follows. " Normally, the dosage is 0.021 mg/kg/week as somatropin (genetical recombination) in 6-7 divided doses by s.c. route. If efficacy is insufficient, the dose may be increased up to 0.47 mg/kg/week in 6-7 divided doses in a week by s.c. route."
  Other Names: Genotropin

SUMMARY:
The objective of this surveillance is to collect information about 1) adverse drug reaction not expected from the LPD (unknown adverse drug reaction), 2) the incidence of adverse drug reactions in this surveillance, and 3)factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Genotropin® should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* Patients need to be administered Somatropin (Genotropin®) in order to be enrolled in the surveillance.

Exclusion Criteria:

* Patients not administered Somatropin (Genotropin®).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A6281292 prescribes the Somatropin (Genotropin® ).
Sampling Method: Probability Sample
Enrollment: 920 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281292&StudyName=Long%20Term%20Use%20of%20Somatropin%20in%20Patients%20Small%20for%20Gestational%20Age

RESULTS

PARTICIPANT FLOW:
Groups:
- Somatropin for Small-for-gestational Age: Participants taking somatropin for small-for-gestational age according to Japanese package insert.
Period: Overall Study
Arm/Group | Somatropin for Small-for-gestational Age
Started | 909
Completed | 890
Not Completed | 19
Not completed — Protocol Violation | 18
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Somatropin for Small-for-gestational Age
Number analyzed (Participants) | 890
Age, Customized [Number; unit: participants]
  <15 years | 884
  >=15 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 423
  Male | 467

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events.
Description: Adverse events mean all unfavorable events that occur in participants after administration of somatropin, irrespective of causal relationship to somatropin (including clinically problematic abnormal changes in laboratory test values). Treatment related adverse events were evaluated in company with the causal relationship to somatropin.
Time Frame: Up to 3 years
Population: The safety analysis population consists of the participants who satisfy the case conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Arm/Group | Somatropin for Small-for-gestational Age
Number analyzed (Participants) | 890
participants | 44

2. Primary Outcome: Number of Unlisted Treatment Related Adverse Events According to Japanese Package Insert.
Description: Adverse events mean all unfavorable events that occur in participants after administration of somatropin, irrespective of causal relationship to somatropin (including clinically problematic abnormal changes in laboratory test values). Treatment related adverse events were evaluated in company with the causal relationship to somatropin. Unlisted treatment related adverse events were confirmed with listed adverse drug reaction according to Japanese package insert.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Somatropin for Small-for-gestational Age
Number analyzed (Participants) | 890
events | 26

3. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin: <15 Years of Age vs. >=15 Years of Age.
Description: To determine whether age is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- <15 Years: Participants younger than 15 years of age when taking somatropin for SGA according to Japanese package insert.
- >=15 Years: Participants 15 years of age or older when taking somatropin for SGA according to Japanese package insert.
Arm/Group | <15 Years | >=15 Years
Number analyzed (Participants) | 884 | 6
participants | 44 | 0
Statistical Analysis 1: Comparison: <15 Years vs >=15 Years; The risk factor tested was "Age". The null hypothesis is that there is no difference between "<15 years and >=15 years" in the frequency of treatment related adverse events; Test type: Superiority or Other; p = 0.575, Chi-squared

4. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin by Gender.
Description: To determine whether gender is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Male: Male Participants taking somatropin for SGA according to Japanese package insert.
- Female: Female Participants taking somatropin for SGA according to Japanese package insert.
Arm/Group | Male | Female
Number analyzed (Participants) | 467 | 423
participants | 19 | 25
Statistical Analysis 1: Comparison: Male vs Female; The risk factor tested was "Gender". The null hypothesis is that there is no difference between "Male and Female" in the frequency of treatment related adverse events; Test type: Superiority or Other; p = 0.206, Chi-squared

5. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin Based on SGA Severity.
Description: To determine whether severity of SGA is a significant risk factor in the frequency of treatment related adverse events. The severity of SGA was comprehensively evaluated on the basis of information including height and weight at birth and height measured one year before the start of administration.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Mild SGA: Participants with mild SGA taking somatropin for SGA according to Japanese package insert.
- Moderate SGA: Participants with moderate SGA taking somatropin for SGA according to Japanese package insert.
- Severe SGA: Participants with severe SGA taking somatropin for SGA according to Japanese package insert.
Arm/Group | Mild SGA | Moderate SGA | Severe SGA
Number analyzed (Participants) | 180 | 479 | 230
participants | 10 | 16 | 18
Statistical Analysis 1: Comparison: Mild SGA vs Moderate SGA vs Severe SGA; The risk factor tested was "Severity". The null hypothesis is that there is no association between "mild, moderate and severe" in the frequency of treatment related adverse events"; Test type: Superiority or Other; p = 0.033, Chi-squared
Statistical Analysis 2: Comparison: Mild SGA vs Moderate SGA vs Severe SGA; "The risk factor tested was "Severity". The null hypothesis is that there is no linear trend in the frequency of treatment related adverse events across increasing levels of severity; Test type: Superiority or Other; p = 0.207, Cochran-Armitage Exact

6. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin: With Past History of Any Disease vs. Without Past History of Any Disease.
Description: To determine whether past history of any disease is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Participants With Past History of Any Disease: Participants with past history of any disease taking somatropin for SGA according to Japanese package insert.
- Participants Without Past History of Any Disease: Participants without past history of any disease taking somatropin for SGA according to Japanese package insert.
Arm/Group | Participants With Past History of Any Disease | Participants Without Past History of Any Disease
Number analyzed (Participants) | 223 | 667
participants | 18 | 26
Statistical Analysis 1: Comparison: Participants With Past History of Any Disease vs Participants Without Past History of Any Disease; The risk factor tested was "Past history of any disease". The null hypothesis is that there is no difference between "With past history of any disease and Without past history any disease" in the frequency of treatment related adverse events; Test type: Superiority or Other; p = 0.013, Chi-squared

7. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin: With Complications vs. Without Complications
Description: To determine whether having complication(s) is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Participants With Complication(s): Participants with complication(s) while taking somatropin for SGA according to Japanese package insert.
- Participants Without Complication(s): Participants without complications while taking somatropin for SGA according to Japanese package insert.
Arm/Group | Participants With Complication(s) | Participants Without Complication(s)
Number analyzed (Participants) | 268 | 622
participants | 21 | 23
Statistical Analysis 1: Comparison: Participants With Complication(s) vs Participants Without Complication(s); The risk factor tested was "Complication(s)". The null hypothesis is that there is no difference between "With complication(s) and Without complication(s)"in the frequency of treatment related adverse events"; Test type: Superiority or Other; p = 0.009, Chi-squared

8. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin: With Hepatic Function Disorder vs. Without Hepatic Function Disorder.
Description: To determine whether hepatic function disorder is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Participants With Hepatic Function Disorder: Participants with hepatic function disorder taking somatropin for SGA according to Japanese package insert.
- Participants Without Hepatic Function Disorder: Participants without hepatic function disorder taking somatropin for SGA according to Japanese package insert.
Arm/Group | Participants With Hepatic Function Disorder | Participants Without Hepatic Function Disorder
Number analyzed (Participants) | 4 | 879
Participants | 3 | 40
Statistical Analysis 1: Comparison: Participants With Hepatic Function Disorder vs Participants Without Hepatic Function Disorder; The risk factor tested was "Hepatic Function Disorder". The null hypothesis is that there is no difference between "with Hepatic Function Disorder and without Hepatic Function Disorder" in the frequency of treatment related adverse events; Test type: Superiority or Other; p < 0.001, Chi-squared

9. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin: With Renal Impairment vs. Without Renal Impairment.
Description: To determine whether renal impairment is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Participants With Renal Impairment: Participants with renal impairment taking somatropin for SGA according to Japanese package insert.
- Participants Without Renal Impairment: Participants without renal impairment taking somatropin for SGA according to Japanese package insert.
Arm/Group | Participants With Renal Impairment | Participants Without Renal Impairment
Number analyzed (Participants) | 9 | 874
Participants | 3 | 40
Statistical Analysis 1: Comparison: Participants With Renal Impairment vs Participants Without Renal Impairment; The risk factor tested was "Renal Impairment". The null hypothesis is that there is no difference between "With Renal Impairment and Without Renal Impairment" in the frequency of treatment related adverse events; Test type: Superiority or Other; p < 0.001, Chi-squared

10. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin: With Concomitant Drug(s) vs. Without Concomitant Drug(s).
Description: To determine whether taking concomitant drug(s) is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Participants With Concomitant Drug(s): Participants taking concomitant drug(s) while taking somatropin for SGA according to Japanese package insert.
- Participants Without Concomitant Drug(s): Participants taking no concomitant drugs while taking somatropin for SGA according to Japanese package insert.
Arm/Group | Participants With Concomitant Drug(s) | Participants Without Concomitant Drug(s)
Number analyzed (Participants) | 250 | 640
Participants | 21 | 23
Statistical Analysis 1: Comparison: Participants With Concomitant Drug(s) vs Participants Without Concomitant Drug(s); The risk factor tested was "Concomitant Drug(s)". The null hypothesis is that there is no difference between "With Concomitant Drug(s) and Without Concomitant Drug(s)" in the frequency of treatment related adverse events; Test type: Superiority or Other; p = 0.003, Chi-squared

11. Primary Outcome: Change in the Growth Rate Standard Deviation (SD) Score for Calendar Age.
Description: Growth rate SD score = (Growth rate - Average growth rate for calendar age of gender) / SD score for growth rate for each calendar age of gender). An SD score indicates how far a participant's score deviates from the mean of the reference population; an SD score higher than the mean gives a positive SD score whereas an SD score lower than the mean gives a negative SD score. In addition, when the bone age was described, it was to be read as the calendar age for men who were 11 years or older and women who were 9 years or older, as necessary.
Time Frame: Up to 3 years
Population: The efficacy analysis population basically consists of the evaluable participants in whom the changes in the growth rate SD score for calendar age and in the height SD score for calendar age were assessed.
Measure: Mean (Standard Deviation); unit: standard deviation (SD) score
Groups:
- Somatropin for Small-for-gestational Age: Participants whose change in the growth rate SD scores was measured at one, two, and three years of taking somatropin for small-for-gestational age according to Japanese package insert.
Arm/Group | Somatropin for Small-for-gestational Age
Number analyzed (Participants) | 855
standard deviation (SD) score
  At one year | 3.9 (2.60)
  At two years | 3.1 (2.54)
  At three years | 2.9 (3.03)
Statistical Analysis 1: Comparison: Somatropin for Small-for-gestational Age; The null hypothesis is that there is no difference in the mean value of the change in the growth rate SD score for calendar age between SGA at one year and SGA at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the hypothesis
Statistical Analysis 2: Comparison: Somatropin for Small-for-gestational Age; The null hypothesis is that there is no difference in the mean value of the change in the growth rate SD score for calendar age between SGA at two years and SGA at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the null hypothesis
Statistical Analysis 3: Comparison: Somatropin for Small-for-gestational Age; The null hypothesis is that there is no difference in the mean value of the change in the growth rate SD score for calendar age between SGA at three years and SGA at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the null hypothesis

12. Primary Outcome: Change in Height SD Score for Calendar Age.
Description: The change in height standard SD for calendar age = (Height SD score for each calendar age - Height SD score for calendar age of the previous year) / (the date on which the height was measured - the date of the previous year on which the height was measured) × 365.25.
Time Frame: Up to 3 years
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: standard deviation (SD) score
Groups:
- Somatropin for Small-for-gestational Age: Participants whose change in the height SD scores was measured at one, two, and three years of taking somatropin for small-for-gestational age according to Japanese package insert.
Arm/Group | Somatropin for Small-for-gestational Age
Number analyzed (Participants) | 855
standard deviation (SD) score
  At one year | 0.6 (0.49)
  At two years | 0.3 (0.41)
  At three years | 0.3 (0.40)
Statistical Analysis 1: Comparison: Somatropin for Small-for-gestational Age; The null hypothesis is that there is no difference in the mean value of the change in the height SD score for calendar age between SGA at one year and SGA at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the null hypothesis
Statistical Analysis 2: Comparison: Somatropin for Small-for-gestational Age; The null hypothesis is that there is no difference in the mean value of the change in the height SD score for calendar age between SGA at two years and SGA at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the null hypothesis
Statistical Analysis 3: Comparison: Somatropin for Small-for-gestational Age; The null hypothesis is that there is no difference in the mean value of the change in the height SD score for calendar age between SGA at three years and SGA at baseline; Test type: Superiority or Other; p < 0.001, t-test, 1 sided; A one-sided paired t-test was performed to test the hypothesis

ADVERSE EVENTS:
Description: The frequency of treatment related adverse events.
Arm/Group | Somatropin for Small-for-gestational Age
Serious Adverse Events (participants affected / at risk) | 8/890
Other Adverse Events (participants affected / at risk) | 36/890
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatropin for Small-for-gestational Age (N=890)
Febrile convulsion (Nervous system disorders) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatropin for Small-for-gestational Age (N=890)
Hypothyroidism (Endocrine disorders) | 2 (2)
Precocious puberty (Endocrine disorders) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperinsulinaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Polydipsia (Metabolism and nutrition disorders) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Pallor (Vascular disorders) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pigmentation lip (Gastrointestinal disorders) | 1 (1)
Malocclusion (Gastrointestinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 2 (2)
Injection site pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Insulin-like growth factor (Investigations) | 1 (1)
Insulin-like growth factor increased (Investigations) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3)
Blood glucose increased (Investigations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Thyroxine free decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.